CLINICAL TRIAL: NCT05647590
Title: SBRT/RT to All Sites of Disease After Three Months of First-line Systemic Chemotherapy in Oligometastatic Stage IV NSCLC Before Maintenance
Brief Title: SBRT/RT in Oligometastatic Stage IV NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ONK-RT+SBRT/CHT
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; radiotherapy; stereotactic robotic radiotherapy; chemotherapy; CyberKnife; acceptable toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Radiotherapy; Maintenance Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSCLC patients (Experimental): Patients with non-small cell lung cancer (NSCLC) will be enrolled in the study.
  Interventions: Procedure: Chemotherapy; Procedure: Radiotherapy (RT) + Stereotactic Body Ratio Therapy (SBRT); Procedure: Maintenance chemotherapy

INTERVENTIONS:
Procedure: Chemotherapy — 3 months of platinum doublet chemotherapy (cDDP / CBDCA + Pemetrexed, NVB)
Procedure: Radiotherapy (RT) + Stereotactic Body Ratio Therapy (SBRT) — * RT to primary tumor + SBRT to all oligometa (max. 10 intra / extracranial lesions, intracranial SD / PR)
  * SBRT V < 100 ml, if technically possible fractionation RT (40 - 50 Gy / 16 - 20 fractions), SBRT (30 Gy / 1 fraction, 50 - 60 Gy / 3 - 5 fractions) 3 - 6 weeks … maintenance
Procedure: Maintenance chemotherapy — Maintenance chemotherapy will follow 3-6 weeks after RT.

SUMMARY:
The core hypothesis to be tested is that the use of consolidative SBRT followed by maintenance chemotherapy in patients with less than or equal to 10 metastatic sites will improve progression-free survival (PFS) with acceptable toxicity compared to maintenance chemotherapy alone.

DETAILED DESCRIPTION:
Lung cancer is the main cause of death from cancer in the Czech Republic and in the world. Non-small cell lung cancer (NSCLC) accounts for more than 80% of all cancer types. Lung cancer is the cause of almost five and a half thousand deaths a year in the Czech Republic, the mortality/incidence ratio is around 85%. The reason is mainly the late recognition of the tumor only in advanced stages - stage III and IV when long-term control of the disease is a rarity. In patients with advanced-stage NSCLC, chemotherapy prolongs overall survival by less than a year on average, which is still a very disappointing result. Therefore, other treatment approaches are being developed to help change this statistic. Radiotherapy (RT) also plays an important role in the treatment of lung cancer, which has a proven therapeutic benefit in both radical and palliative indications for up to 76% of all patients.

Stereotactic Robotic Radiotherapy (SBRT) achieves extraordinary precision due to the precise definition of the target volume with maximum sparing of surrounding tissues. It also allows you to focus on bearings that show movement, especially during the breathing cycle. Radiotherapy, whether conventional or stereotactic, is a non-invasive treatment method.

The aim of the study is to verify the feasibility of consolidation SBRT - CyberKnife with subsequent maintenance chemotherapy in patients in IV. The stage of non-small cell lung cancer with a maximum of 10 metastatic foci, with acceptable toxicity, while maintaining a good quality of life. The time to progression (worsening of the disease), overall survival, the number of foci with local control, the time to the appearance of new foci, the duration of maintenance chemotherapy, and the finding of predictive molecular markers of treatment response will be evaluated.

Design: prospective, interventional trial (University Hospital Ostrava) 3 months of chemotherapy platin doublet (cDDP / CBDCA + Pemetrexed, NVB) if SD/PD: RT to primary tumour + SBRT to all oligometa (max. 10 intra / extrarnial leasions, intracranial SD / PR) SBRT V < 100 ml, if technically possible fractionation RT (40 - 50 Gy / 16 - 20 fractions), SBRT (30 Gy / 1 fraction, 50 - 60 Gy / 3 - 5 fractions) 3 - 6 weeks … maintenance

Preliminary examination: PET/CT, ECHO, spirometry, MR (only if neurological symptomatology)

Endpoints:

Primary Endpoints: toxicity (CTCAE ver. 4), PFS Secondary Endpoints: OS, local control, time to new lesion, duration of maintenance chemotherapy, restriction volume according to spirometry, EF

Ad hoc analysis: PDL1 expression, Ki67 status, smoking history, KPS

Restage: every three 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven metastatic NSCLC (Stage IV).
* Patients must have received three months of first-line chemotherapy and achieved stable disease or partial response.
* Age ≥ 18 years
* Patients must have measurable disease at baseline.
* Patients can have up to 10 discrete active extracranial/intracranial lesions identified by PET/CT or MRI scan within 8 weeks prior to the initiation of SBRT.
* Patients must have a Karnofsky Performance Scale (KPS) >60
* AST, ALT & Alkaline phosphates must be ≤ 2.5x the upper limit of normal. Total bilirubin must be within the limit of normal.
* Patients should have adequate bone marrow function as defined by peripheral granulocyte count of ≥1500/mm³.
* Patients should have adequate renal function (serum creatinine ≤1.5 times the upper limit of normal (ULN).
* Females of childbearing potential should have a negative pregnancy test.
* Patients who would be receiving SBRT for lung tumors must have a documented forced expiratory volume in 1 second (FEV1) ≥ 1L.
* Patients must provide verbal and written informed consent to participate in the study

Exclusion Criteria:

* Patients receiving first-line erlotinib, gefitinib, or crizotinib for EGFR mutant-positive or EML4-ALK-positive NSCLC will be excluded.
* Patients who previously received radiotherapy at the primary site with CT evidence of disease progression at the primary site within 3 months following the initial radiotherapy
* Patients with serious, uncontrolled, concurrent infection(s)
* Significant weight loss (>10%) in the prior 3 months
* Patients with cutaneous metastasis of NSCLC
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cancers
* Patients with more than 10 discrete extra/intracranial lesions
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Patients who are pregnant; patients with reproductive capability will need to use adequate contraception during the time of participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Grade of Toxicity | up to 12 months
  Grade of toxicity of the treatment will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4
Progression-Free Survival | up to 12 months
  Progression-free survival (PFS) will be observed (in months)

SECONDARY OUTCOMES:
Overall Survival | up to 12 months
  Overall survival (OS) will be observed (in months)
Time to new lesion | up to 12 months)
  Time to new lesion will be observed (in months)
Duration of maintenance chemotherapy | up to 12 months
  Duration of maintenance chemotherapy will be observed (in months)
Restriction volume of pulmonary capacity | up to 12 months
  The restriction volume of pulmonary capacity (in %, compared to the vital capacity and total lung capacity)

CONTACTS AND LOCATIONS:
Overall Officials: Tereza Paračková, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.